CLINICAL TRIAL: NCT01297764
Title: A Phase I/II Study of Carfilzomib, Lenalidomide, Vorinostat, and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Carfilzomib, Lenalidomide, Vorinostat, and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Acronym: QUAD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002074 - QUAD RV-0549
Record Dates: First submitted 2011-02-11; First posted 2011-02-17 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat; Lenalidomide; carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carfilzomib for MML (Experimental): Vorinostat, Lenalidomide, Carfilzomib, Dexamethasone - This study will be conducted as an open-label Phase I/II, single-center study in which subjects will receive carfilzomib, lenalidomide, vorinostat and dexamethasone, for relapsed and/or refractory multiple myeloma. Study treatment will be administered in sequential cohorts, with 3-6 subjects in each cohort. Treatment will be administered in 28-day cycles, with the fourth week as a rest week, for 12 cycles or until disease progression or unacceptable toxicity develops.
  Interventions: Drug: Vorinostat, Lenalidomide, Carfilzomib, Dexamethasone

INTERVENTIONS:
Drug: Vorinostat, Lenalidomide, Carfilzomib, Dexamethasone — Dose Escalation Schema Cohort Carfilzomib (mg/m2) Lenalidomide (mg) Vorinostat (mg) Dexamethasone (mg)
  1. 15 15 300 40
  2. 20 15 300 40
  3. 20 25 300 40
  4. 20/27* 25 300 40
  5. 20/27* 25 400 40
  Other Names: Vorinostat (Zolinza); Lenalidomide (Revlimid); Carfilzomib (Kyprolis); Dexamethasone (Decadron, Baycadron)

SUMMARY:
This study will evaluate the feasibility of combining four of the most active agents available for the treatment of multiple myeloma. Further the investigators will attempt to assess the activity of this combination.

DETAILED DESCRIPTION:
Phase I/II studies of the novel proteasome inhibitor, carfilzomib, have shown it to have significant activity in patients with advanced multiple myeloma, including patients with bortezomib refractory disease. This drug, unlike bortezomib, has minimal neurotoxicity and appears to have minimal gastrointestinal (GI) toxicity. Experience with the combination of bortezomib, lenalidomide and dexamethasone has shown both neuropathy and chronic diarrhea to be limiting.

Vorinostat is a histone deacetylase inhibitor with modest single agent activity in multiple myeloma. Dysesthesia, GI issues and fatigue have been problematic in this patient population. More recent studies combining vorinostat with lenalidomide and dexamethasone or with bortezomib have demonstrated a much more robust activity, including in patients refractory to lenalidomide or bortezomib-based combinations. Again, neuropathy, fatigue and GI issues have been problematic.

The investigators own anecdotal experience with combinations of proteasome inhibitor, histone deacetylase inhibitor, immunomodulators and dexamethasone has shown this combination to be extremely active and well tolerated. The combination of vorinostat, carfilzomib, lenalidomide and dexamethasone should offer the opportunity to maximize activity while limiting toxicities, particularly neuropathy and GI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible to enroll in this study:

Disease related:

1. Symptomatic multiple myeloma
2. Relapsed and/or refractory multiple myeloma after at least one prior therapeutic regimen for multiple myeloma
3. Prior treatment with immunomodulatory agents, proteasome inhibitors and histone deacetylase inhibitors is permitted. (Patients who have used HDAC inhibitors, including valproic acid , must have at least 5 half-lives wash out period before beginning therapy with vorinostat on this protocol.)
4. Measurable disease, as indicated by one or more of the following:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine Bence-Jones protein ≥ 200 mg/24 h
   * If Serum Protein Electrophoresis is felt to be unreliable for routine M-protein measurement (particularly for patients with IgA MM), then quantitative immunoglobulin levels can be accepted.
   * Serum free light chain ≥ 10 mg/dL (≥ 100 mg/L) and an abnormal free light chain ratio

   Demographic
5. Males and females ≥ 18 years of age
6. Life expectancy of more than three months
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 (see Appendix B)

Laboratory

8.Adequate hepatic function, with bilirubin < 2 times the upper limit of normal (ULN) and alanine aminotransferase (ALT) < 3 times ULN 9.Absolute neutrophil count (ANC) ≥ 1,000/mm3 Hemoglobin ≥ 8 gm/dL Platelet count ≥ 50,000/ mm3 (≥ 30 × 109/L if myeloma involvement in the bone marrow is > 50%)

* Screening ANC should be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G CSF for at least 2 weeks.
* Subjects may receive red blood cell (RBC) or platelet transfusions, if clinically indicated, in accordance with institutional guidelines
* Screening platelet count should be independent of platelet transfusions for at least 2 weeks 10.Calculated or measured creatinine clearance of ≥60 mL/minute, calculated using the formula of Cockcroft and Gault [(140 - Age) x Mass (kg) / (72 x creatinine mg/dL)]; multiply result by 0.85 (if female). Other generally accepted calculation methods can be substituted.11.Potassium level 3.5-5.2 meq/L (institutional normal range) Ethical/Other 12.Written informed consent in accordance with federal, local, and institutional guidelines 13.Females of Child Bearing Potential* (FCBP) must have a negative serum or urine pregnancy test, with a sensitivity of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescription must be filled with 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO methods of acceptable methods of birth control, one highly effective method AND one additional effective method of birth control (contraception) AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy Testing. (See Appendix G: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods)

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

    14. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy (See Appendix G: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods) 15. All study participants must be registered into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist®.

    16. Subjects must adhere to the study visit schedule and other protocol requirements and receive outpatient treatment and laboratory monitoring at the institute that administers the drug 17. Subjects must agree to take enteric-coated aspirin 81-325 mg orally daily, or if history of prior thrombotic disease or allergy to aspirin, must be fully anticoagulated with warfarin (INR 2-3) or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism.

Exclusion Criteria

Subjects who meet any of the following exclusion criteria are not eligible to be enrolled in this study:

Disease related

1. Subjects with non-secretory or hyposecretory multiple myeloma, defined as <0.5 g/dL M-protein in serum and <200 mg/24 hr Bence Jones protein in urine and serum free light chain <10mg/dL (<100 mg/L) and no measurable plasmacytoma
2. Corticosteroid therapy in a dose equivalent to dexamethasone ≥ 4 mg/day or prednisone ≥20 mg/day within 3 weeks prior to first dose
3. Concurrent use of histone deacetylase inhibitor (eg. Valproic acid)
4. Use of any other experimental drug or therapy within 28 days of baseline
5. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
6. Waldenström's macroglobulinemia
7. Chemotherapy with approved or investigative anticancer therapeutics, including steroid therapy dose as defined above, within 2 weeks prior to first dose
8. Radiation therapy within 1 week prior to first dose, Immunotherapy within 3 weeks prior to first dose . Planned radiation therapy that occurs after the start of treatment
9. Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater.

   Concurrent conditions
10. Pregnant or lactating females (Lactating females must agree not to breast feed while taking lenalidomide or vorinostat).
11. History of allergy to boron or mannitol
12. Major surgery within 2 weeks prior to first dose
13. Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction in the previous six months
14. Uncontrolled hypertension
15. Acute active infection requiring intravenous antibiotics, antivirals, or antifungals within one week prior to first dose or oral antibiotics within 1 week
16. Known or suspected HIV infection, known HIV seropositivity, or active hepatitis A, B, or C infection.
17. Serious psychiatric or medical conditions that could interfere with treatment
18. Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment
19. Contraindication to any of the required concomitant drugs, including proton-pump inhibitor (e.g., lansoprazole), antiviral agents, enteric-coated aspirin or other anticoagulant, or if a history of prior thrombotic disease, warfarin or low molecular weight heparin
20. Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment
21. Subjects with pleural effusions requiring therapeutic thoracentesis or ascites requiring therapeutic paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety and dose of carfilzomib, lenalidomide, vorinostat and dexamethasone for MM | Within 30 days of the last administration of study treatment
  Primary Objective: To evaluate safety and establish the maximum tolerated dose (MTD) [and/or a protocol defined dose below the MTD] of carfilzomib, lenalidomide, vorinostat and dexamethasone in relapsed and/or refractory multiple myeloma subjects.
  Secondary Objectives: To observe evidence of efficacy (response rate, duration of response, time to progression, time to next treatment)

SECONDARY OUTCOMES:
Overall response rate (ORR) Time to next treatment (TTNT) Time to progression (TTP) Duration of response (DOR | Within 30 days of the last administration of study treatment
  Secondary Objectives: To observe evidence of efficacy (response rate, duration of response, time to progression, time to next treatment)

CONTACTS AND LOCATIONS:
Overall Officials: David Siegel, MD, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Ries LAG, Melbert D, Krapcho M, Mariotto A, Miller BA, Feuer EJ, et al (eds). SEER Cancer Statistics Review, 1975-2004, National Cancer Institute. Bethesda, MD, http://seer.cancer.gov/csr/1975_2004/, based on November 2006 SEER data submission, posted to the SEER website, 2007.
- [Background] Jawed I, Lee CM, Tward JD, Macdonald OK, Martincic D, Vudarla N, Fairbanks RK, et al. Survival outcomes for multiple myeloma over three decades: a surveillance, epidemiology, and end results (SEER) analysis. J Clin Oncol. 2007 ASCO Annual Meeting Proceedings Part I. Vol 25, No. 18S (June 20 Supplement), 2007:8019.
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Richardson PG, Jagannath S, Avigan DE, Alsina M, Schlossman RL, Mazumder A, et al. Lenalidomide plus bortezomib (Rev-Vel) in relapsed and/or refractory multiple myeloma (MM): final results of a multicenter phase 1 trial. Blood. 2006 Nov 16;108(11):Abstract #405.
- [Background] Richardson P, Schlossman RL, Mitsiades CS, Munshi NC, Colson K, Doss D, et al. Phase I clinical trial of oral administration of the histone deacetylase (HDAC) inhibitor suberoylanilide hydroxamic acid (SAHA) in patients with relapsed/refractory multiple myeloma (MM). [Abstract]. Blood 2004;104(11):420a.
- [Background] Mitsiades N, Mitsiades CS, Richardson PG, McMullan C, Poulaki V, Fanourakis G, Schlossman R, Chauhan D, Munshi NC, Hideshima T, Richon VM, Marks PA, Anderson KC. Molecular sequelae of histone deacetylase inhibition in human malignant B cells. Blood. 2003 May 15;101(10):4055-62. doi: 10.1182/blood-2002-11-3514. Epub 2003 Jan 16. PMID 12531799
- [Background] Mitsiades CS, Mitsiades NS, McMullan CJ, Poulaki V, Shringarpure R, Hideshima T, Akiyama M, Chauhan D, Munshi N, Gu X, Bailey C, Joseph M, Libermann TA, Richon VM, Marks PA, Anderson KC. Transcriptional signature of histone deacetylase inhibition in multiple myeloma: biological and clinical implications. Proc Natl Acad Sci U S A. 2004 Jan 13;101(2):540-5. doi: 10.1073/pnas.2536759100. Epub 2003 Dec 26. PMID 14695887
- [Background] Siegel D, Weber DM, Mitsiades CS, Dimopoulo MA, Harousseau JL, Rizvi S, et al. Combined Vorinostat, Lenalidomide and Dexamethasone Therapy in Patients with Relapsed or Refractory Multiple Myeloma: A Phase I Study. [Abstract] Blood (ASH Annual Meeting Abstracts) 2009;114(22)304a.
- [Background] Pei XY, Dai Y, Grant S. Synergistic induction of oxidative injury and apoptosis in human multiple myeloma cells by the proteasome inhibitor bortezomib and histone deacetylase inhibitors. Clin Cancer Res. 2004 Jun 1;10(11):3839-52. doi: 10.1158/1078-0432.CCR-03-0561. PMID 15173093
- [Background] Prince HM, Bishton M, Harrison S. The potential of histone deacetylase inhibitors for the treatment of multiple myeloma. Leuk Lymphoma. 2008 Mar;49(3):385-7. doi: 10.1080/10428190801950058. PMID 18297514
- [Background] Richardson PG, Mitsiades CS, Colson K, Reilly E, McBride L, Chiao J, et al. Final results of a phase I trial of oral vorinostat (suberoylanilide hydroxamic acid, SAHA) in combination with bortezomib in patients with advanced multiple myeloma [Abstract]. Blood (ASH Annual Meeting Abstracts) 2007;110(11):1179.
- [Background] Weber DM, Jagannath S, Mazumder A, Sobecks R, Schiller GJ, Gavino M, et al. Phase I trial of oral vorinostat (suberoylanilide hydroxamic acid, SAHA) in combination with bortezomib in patients with advanced multiple myeloma [Abstract]. Blood (ASH Annual Meeting Abstracts) 2007;110(11):1172.
- [Background] Weber D, Badros AZ, Jagannath S, Siegel D, Richon V, Rizvi S, Garcia-Vargas J, Reiser D and Anderson KC. Vorinostat Plus Bortezomib for the Treatment of Relapsed/Refractory Multiple Myeloma (MM): Early Clinical Experience. American Society of Hematology Annual Meeting Abstract Nov 2008;112:871.
- [Background] Badros A, Philip S, Niesvizky R, Goloubeva O, Harris C, Zwiebel J, et al. Phase I trial of vorinostat (suberoylanilide hydroxamic acid, SAHA) plus bortezomib (Bort) in relapsed and refractory multiple myeloma (MM) patients (pts.). EHA (European Hematology Association annual Meeting Abstracts) 2008;93(s1)0642:258
- [Background] Demo SD, Kirk CJ, Aujay MA, Buchholz TJ, Dajee M, Ho MN, Jiang J, Laidig GJ, Lewis ER, Parlati F, Shenk KD, Smyth MS, Sun CM, Vallone MK, Woo TM, Molineaux CJ, Bennett MK. Antitumor activity of PR-171, a novel irreversible inhibitor of the proteasome. Cancer Res. 2007 Jul 1;67(13):6383-91. doi: 10.1158/0008-5472.CAN-06-4086. PMID 17616698
- [Background] Ivancsits D, Nimmanapali R, Sun M, Shenk K, Demo S, Bennett D, et al. The proteasome inhibitor PR-171 inhibits cell growth, induces apoptosis, and overcomes de novo and acquired drug resistance in human multiple myeloma cells. Blood 2006;106:452a.
- [Background] Demo SD, Buchholz TJ, Laidig GL, Parlati F, Shenk KD, Smyth MS, et al. Biochemical and cellular characterization of the novel proteasome inhibitor PR-171. Blood 2006;106:455a.
- [Background] Kuhn DJ, Chen Q, Voorhees PM, Strader JS, Shenk KD, Sun CM, Demo SD, Bennett MK, van Leeuwen FW, Chanan-Khan AA, Orlowski RZ. Potent activity of carfilzomib, a novel, irreversible inhibitor of the ubiquitin-proteasome pathway, against preclinical models of multiple myeloma. Blood. 2007 Nov 1;110(9):3281-90. doi: 10.1182/blood-2007-01-065888. Epub 2007 Jun 25. PMID 17591945
- [Background] Lonial S, Waller EK, Richardson PG, Jagannath S, Orlowski RZ, Giver CR, Jaye DL, Francis D, Giusti S, Torre C, Barlogie B, Berenson JR, Singhal S, Schenkein DP, Esseltine DL, Anderson J, Xiao H, Heffner LT, Anderson KC; SUMMIT/CREST Investigators. Risk factors and kinetics of thrombocytopenia associated with bortezomib for relapsed, refractory multiple myeloma. Blood. 2005 Dec 1;106(12):3777-84. doi: 10.1182/blood-2005-03-1173. Epub 2005 Aug 11. PMID 16099887
- [Background] Stewart KA, O'Connor OA, Alsina M, Trudel S, Urquilla PR, Vallone MK, et al. Phase I evaluation of carfilzomib (PR-171) in hematological malignancies: responses in multiple myeloma and Waldenstrom's macroglobulinemia at well-tolerated doses. J Clin Oncol. 2007 ASCO Annual Meeting Proceedings Part I. Vol 25, No. 18S (June 20 Supplement), 2007: 8003.
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033